CLINICAL TRIAL: NCT06455501
Title: FOAM: Functional Outcome After Ventral Mesh Rectopexy, Prospective Cohort Study
Brief Title: FOAM: Functional Outcome After Ventral Mesh Rectopexy
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: FOAM-trial
Record Dates: First submitted 2024-05-15; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Rectal Prolapse
Keywords: Ventral mesh rectopexy; Laparoscopic ventral mesh rectopexy; Quality of Life; Bowel function; Recurrence; Sexual function
MeSH Terms: conditions — Rectal Prolapse; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ventral mesh rectopexy — Ventral mesh rectopexy is performed with a superficial peritoneal incision from the right side of the sacral promontory, extended over the right outer border of the mesorectum, towards the deepest part of pouch of Douglas, sparing the right hypogastric nerve. In women, the vagina is retracted anteriorly and a dissection of the rectovaginal septum is performed down to the pelvic floor. A strip of mesh is attached to the ventral part of distal rectum and then fixed upon the sacral promontory.

SUMMARY:
Rectal prolapse is a protrusion of rectal wall through the anus. A surgical technique called Ventral mesh rectopexy has become a standard procedure for this condition in many centers.

The goal of this trial is to investigate functional outcome, recurrence rates and complications after ventral mesh rectopexy. The main question it aims to answer is:

- Do bowel function, quality of life and sexual function improve after Ventral mesh rectopexy?

Participants will:

* be asked to fill in questionaires before surgery, 3-6 months after surgery and 12 months after surgery.
* be examined by a surgeon 3-6 months, 12 months and 3 years after surgery.

DETAILED DESCRIPTION:
Several different procedures have been described for surgical treatment of rectal prolapse and a consensus has not yet been reached. Over the past 20 years, the use of Ventral mesh rectopexy to treat external rectal prolapse has gained increasing worldwide acceptance. Ventral mesh rectopexy has become a standard procedure in many centers based on low recurrence rates, limited complications and good functional results but the use and type of mesh have been debated. Concerns have also been expressed regarding the choice of surgical technique, which differs between centers, and the lack of high-level evidence.

There are few prospective trials and the use of LVMR in a Swedish setting has not yet been evaluated. FOAM (Functional Outcome After ventral Mesh rectopexy) therefore aims to investigate bowel function, quality of life, sexual function, recurrence rates and complications after ventral mesh rectopexy.

A prospective cohort study on patients undergoing ventral mesh rectopexy for external rectal prolapse in Sweden will be conducted. Approximately 70 patients will be included at a maximum of 10 hospitals in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* full-thickness rectal prolapse
* the surgeon agrees that ventral mesh rectopexy is needed for the condition
* capable of participating in follow-up visits and answering questionnaires
* informed consent

Exclusion Criteria:

* patient below 18 years of age
* ongoing pregnancy
* inability to understand the Swedish language
* dementia or other cognitive disorder that unables informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing ventral mesh rectopexy for full-thickness rectal prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Bowel function | Evaluated at baseline, 3-6 months and 12 months postoperatively
  Wexner constipation score: scale 0-30, 30=worst outcome
Bowel function | Evaluated at baseline, 3-6 months and 12 months postoperatively
  Wexner incontinence score: scale 0-20, 20=worst outcome
Bowel function | Evaluated at baseline, 3-6 months and 12 months postoperatively
  Colo-rectal-anal Distress Inventory (CRADI-8): scale 0-100 (100=worst outcome)
Quality of Life after surgery | Evaluated at baseline, 3-6 months and 12 months postoperatively
  Colorectal-Anal Impact Questionnaire (CRAIQ-7): scale 0-100, 100=worst outcome
Sexual function | Evaluated at baseline, 3-6 months and 12 months postoperatively
  PROMIS Sexual function and satisfaction version 2.0. Selected domains: Interest in sexual activity (scale 2-10, 10=highest interest), sexual activity screener (scale yes/no) and satisfaction with sex life (scale 2-10, 10=highest satisfaction)

SECONDARY OUTCOMES:
Recurrence rate | Evaluated at baseline, 3-6 months, 12 months and 3 years postoperatively. Clinical examination by surgeon will be performed to evaluate recurrence.
  Recurrence of rectal prolapse
Postoperative complications | Within 30 days postoperatively
  Clavien Dindo classification
Long-term complications | Evaluated at baseline, 3-6 months, 12 months and 3 years postoperatively.
  Ileus, pelvic abscess, mesh erosion, other complications
Length of stay | From day of operation to day of discharge from hospital, reported at follow-up 3-6 months postoperatively.
  Stay in hospital postoperatively
Mortality | Within 30 days postoperatively
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Graf, Professor, Principal Investigator — Department of Surgical Sciences, Uppsala Universitet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tou S, Brown SR, Nelson RL. Surgery for complete (full-thickness) rectal prolapse in adults. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD001758. doi: 10.1002/14651858.CD001758.pub3. PMID 26599079
- [Background] D'Hoore A, Cadoni R, Penninckx F. Long-term outcome of laparoscopic ventral rectopexy for total rectal prolapse. Br J Surg. 2004 Nov;91(11):1500-5. doi: 10.1002/bjs.4779. PMID 15499644
- [Background] Badrek-Al Amoudi AH, Greenslade GL, Dixon AR. How to deal with complications after laparoscopic ventral mesh rectopexy: lessons learnt from a tertiary referral centre. Colorectal Dis. 2013 Jun;15(6):707-12. doi: 10.1111/codi.12164. PMID 23384148
- [Background] Evans C, Stevenson AR, Sileri P, Mercer-Jones MA, Dixon AR, Cunningham C, Jones OM, Lindsey I. A Multicenter Collaboration to Assess the Safety of Laparoscopic Ventral Rectopexy. Dis Colon Rectum. 2015 Aug;58(8):799-807. doi: 10.1097/DCR.0000000000000402. PMID 26163960
- [Background] Randall J, Smyth E, McCarthy K, Dixon AR. Outcome of laparoscopic ventral mesh rectopexy for external rectal prolapse. Colorectal Dis. 2014 Nov;16(11):914-9. doi: 10.1111/codi.12741. PMID 25110205
- [Background] Teleman P, Stenzelius K, Iorizzo L, Jakobsson U. Validation of the Swedish short forms of the Pelvic Floor Impact Questionnaire (PFIQ-7), Pelvic Floor Distress Inventory (PFDI-20) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Acta Obstet Gynecol Scand. 2011 May;90(5):483-7. doi: 10.1111/j.1600-0412.2011.01085.x. PMID 21306343
- [Background] Hoven E, Flynn KE, Weinfurt KP, Eriksson LE, Wettergren L. Psychometric evaluation of the Swedish version of the PROMIS Sexual Function and Satisfaction Measures in clinical and nonclinical young adult populations. Sex Med. 2023 Jan 12;11(1):qfac006. doi: 10.1093/sexmed/qfac006. eCollection 2023 Feb. PMID 37007849
- [Background] Wexner SD. Further validation of the Wexner Incontinence Score: A note of appreciation and gratitude. Surgery. 2021 Jul;170(1):53-54. doi: 10.1016/j.surg.2021.02.039. Epub 2021 Apr 15. No abstract available. PMID 33863582
- [Background] Agachan F, Chen T, Pfeifer J, Reissman P, Wexner SD. A constipation scoring system to simplify evaluation and management of constipated patients. Dis Colon Rectum. 1996 Jun;39(6):681-5. doi: 10.1007/BF02056950. PMID 8646957